CLINICAL TRIAL: NCT04358523
Title: Drug Interaction Between RDV and SOF in ASC18 Tablets (RDV/SOF Compound Tablets) and the Influence of Food Effect on the Pharmacokinetics of ASC18 Tablets Were Evaluated in Healthy Subjects. Comparison of the Pharmacokinetic Parameters of ASC18 Tablets（Ravidasvir and Sofosbuvir Fixed Dose Combination）With Reference Tablets (Ravidasvir Sofosbuvir) in Healthy Subjects After Single and Multiple Oral Dosing
Brief Title: A Study of the Relative Bioavailability of ASC18 Tablets vs Reference Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASC-ASC18-I-CTP-01
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — ravidasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC18 (D1,D4-13）;RDV + SOF(D27,D30-39) (Experimental): ASC18 one tablet (200mg RDV+400mg SOF / tablet) at a time, once per day, day 1 and day 4 to 13. RDV one tablet (200mg / tablet) SOF one tablet (400mg/tablet)at a time, once per day, day 27 and day 30 to 39.
  Interventions: Drug: ASC18; Drug: ravidasvir and sofosbuvir
- RDV + SOF (D1,D4-13）;ASC18(D27,D30-39) (Experimental): RDV one tablet (200mg / tablet) SOF one tablet (400mg/tablet)at a time, once per day, day 1 and day 4 to 13. ASC18 one tablet (200mg RDV+400mg SOF / tablet) at a time, once per day, day 27 and day 30 to 39.
  Interventions: Drug: ravidasvir and sofosbuvir; Drug: ASC18

INTERVENTIONS:
Drug: ASC18 — ASC18：ravidasvir and sofosbuvir fixed Dose Combination 200 mg/400 mg
  Arms: ASC18 (D1,D4-13）;RDV + SOF(D27,D30-39)
Drug: ravidasvir and sofosbuvir — RDV 200 mg and SOF 400 mg
Drug: ASC18 — ASC18：ravidasvir and sofosbuvir fixed Dose Combination 200 mg/400 mg
  Arms: RDV + SOF (D1,D4-13）;ASC18(D27,D30-39)

SUMMARY:
The objective of this study is to evaluate potential drug interaction between RDV and SOF in ASC18 tablets (RDV/SOF compound tablets) and the influence of food effect on the pharmacokinetics of ASC18 tablets were evaluated in healthy subjects -and compare the pharmacokinetic parameters of ASC18 tablets（ravidasvir and sofosbuvir fixed dose combination）with ravidasvir tablets and sofosbuvir tablets in healthy subjects after single and multiple oral dosing.

DETAILED DESCRIPTION:
This randomized, open-label, crossover study will evaluate the relative bioavailability of ASC18 (ravidasvir and sofosbuvir fixed dose combination) tablets as compared to ad hoc combination of reference tablets of ravidasvir and sofosbuvir in healthy volunteers. Subjects will be randomized to 1 of 2 treatment sequences to receive multiple oral doses of either ASC18 tablets (ravidasvir and sofosbuvir fixed Dose Combination) or ravidasvir and sofosbuvir as separate tablets. In the crossover design, subjects will participate in 2 study periods with at least a 14-day washout between periods.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 (including 18 and 45 years old), both male and female.
2. Male body weight ≥ 50 kg, female body weight ≥ 45 kg; BMI between 19-24 kg / m2 (including boundary value).
3. According to the medical history, hearing examination, physical examination, vital signs, laboratory examination and 12 lead electrocardiogram (ECG) examination, the general health condition is good, and there is no clinically significant abnormality in each index.
4. There was no family planning in the past half a year, and they were willing to take effective contraceptive measures within half a year after the last administration.
5. Non pregnant or lactating women.
6. Serum creatinine measured during screening evaluation and creatinine clearance rate (CrCl) from actual body weight (greater than or equal to 80 ml / min (using Cockcroft Gault method)).
7. Voluntary signing of informed consent.

Exclusion Criteria:

* (1) Have or are currently suffering from any serious clinical disease such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormality, or any other disease (such as anemia, hearing impairment, hyperthyroidism, etc.) that can interfere with the test results.

  (2) Family history of malignant tumor, history of epilepsy, history of tuberculosis or contact history of tuberculosis patients.

  (3) Has had gastrointestinal surgery, vagotomy, enterotomy, or any surgery (other than herniorrhaphy, appendectomy) that may interfere with gastrointestinal peristalsis, pH, or absorption.

  (4) Those with drug allergy constitution, including those with drug or food allergy history.

  (5) Any prescription medicine, over-the-counter medicine, any vitamin product or herbal medicine, such as St. John's wort, echinacea, silymarin (i.e. silymarin), Xiaochaihu Decoction, was used within 14 days before the first administration. (6) Smokers or those who smoked more than 5 cigarettes per day in 3 months before the trial.

  (7) Alcoholics or regular drinkers within 6 months before the test, i.e. drinking more than 14 units of alcohol per week (1 unit = 360 ml of beer or 45 ml of spirits with 40% alcohol or 150 ml of wine).

  (8) Those who drink too much tea, coffee or caffeinated beverage (more than 8 cups, 1 cup = 250 ml) every day within 3 months before the first administration. (9) 48 hours before taking the first research, any food or drink containing caffeine or coffee (rich in tea, chocolate, etc.) or foods rich in xanthine (e.g. sardine, animal liver, etc.) or beverage were consumed or planned.

  (10) Blood donation or blood loss of more than 400ml occurred within 3 months before the first administration.

  (11) Those who had participated in other clinical trials and received study drug treatment within 3 months before the first administration.

  (12) Those who have used the oral contraceptive within 30 days before the first administration, or those who have used the long-acting estrogen or progesterone injection or implant within 6 months before the first administration.

  (13) There were unprotected actors (women) within 14 days before the first administration.

  (14) Those who have special requirements for diet and cannot follow the unified diet.

  (15) Subjects who could not tolerate the high fat and high calorie breakfast (this article only applies to the subjects who participated in the PK effect test of food). (16) Irregular defecation within 7 days before the first administration.

  (17) Unqualified alcohol test or positive drug abuse screening. (18) HBsAg, HCV AB, HIV AB and Treponema pallidum were positive. (19) In addition to the above, the researcher judged that it was not suitable to participate in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of ASC18 in healthy volunteers: number of Adverse Events | Up to 93 days
  Evaluate number of Adverse Events as a measure of safety and tolerability of ASC18.

SECONDARY OUTCOMES:
Cmax of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days.
  Evaluate the Peak Plasma Concentration after single and multiple oral doses of ASC18 administered to Chinese healthy volunteers.
Tmax of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days
  Evaluate the Time to reach the maximum plasma concentration after single and multiple oral doses of ASC18 administered to Chinese healthy volunteers.
AUC of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days
  Evaluate the Area under the plasma concentration versus time curve after single and multiple oral doses of ASC18 administered to Chinese healthy volunteers.
t1/2 of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days
  Evaluate the Terminal-Phase Half-Life after single and multiple oral doses of ASC18 administered to Chinese healthy volunteers volunteers.
CL/F of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days
  Evaluate the Apparent Systemic Clearance after single oral dose of ASC18 administered to Chinese healthy volunteers.
Vd/F of ASC18 | On Day 1,2,3 after single doses and On Day 1,2,3,4 after multiple doses, respectively. The entire study will last up to 93 days
  Evaluate the Apparent Volume of Distribution after single oral dose of ASC18 administered to Chinese healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, MD, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided